CLINICAL TRIAL: NCT06925386
Title: The Relationship Between Microbioma Balance and Acne Vulgaris as a New Acne Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: PT. Prodia Stem Cell Indonesia (Industry); B-Crobes Laboratory (M) Sdn Bhd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHAR-202503.01
Record Dates: First submitted 2025-03-20; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Standard of Care; Secretome

STUDY DESIGN:
Intervention Model Description: A parallel group design with four arms was used, (1) standard therapy with oral probiotics and topical secretome (placebo), (2) standard therapy with oral probiotics (placebo) and topical secretome, (3) standard therapy with oral probiotics and topical secretome, and (4) standard therapy with oral probiotics (placebo) and topical secretome (placebo). Participants were assigned to groups using a random permuted block sampling method (comprising A, B, C, D). This method is commonly applied in clinical trials including small sample sizes with staggered participants' enrollment. Observation spans 8 weeks. All groups were subjected to pretest and posttest assessments, measuring acne severity, fecal microbiome metabolites, skin condition, and IL-6 before and after intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Standard therapy + oral probiotics + topical secretome (placebo)
  Interventions: Drug: Standard therapy; Dietary Supplement: HEXBIO
- Group 2 (Experimental): Standard therapy + oral probiotics (placebo) + topical secretome
  Interventions: Drug: Standard therapy; Biological: Secretome
- Group 3 (Experimental): Standard therapy + oral probiotics + topical secretome
  Interventions: Drug: Standard therapy; Dietary Supplement: HEXBIO; Biological: Secretome
- Group 4 (Placebo Comparator): Standard therapy + oral probiotics (placebo) + topical secretome (placebo)
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Standard therapy — The standard therapy for participants included a structured skincare regimen. A face wash was used once daily before bedtime to cleanse the skin. In the morning, a non-comedogenic sunscreen and a moisturizer were applied to protect and hydrate the skin. Additionally, a night cream containing clindamycin and tretinoin was applied once daily at night, specifically on acne-affected areas, to target inflammation and promote skin renewal.
Dietary Supplement: HEXBIO — The oral probiotics given are Hexbio®, an oral probiotic containing multiple beneficial bacterial strains, including Lactobacillus acidophilus BCMC® 12130, Lactobacillus casei BCMC® 12313, Lactobacillus lactis BCMC® 12451, Bifidobacterium bifidum BCMC®02290, Bifidobacterium longum BCMC® 02120, and Bifidobacterium infantis BCMC®02129. This probiotic was administered in granule form and swallowed directly. Participants consumed the probiotic twice daily, after breakfast and dinner, for eight weeks to support gut microbiome balance and potential skin health benefits.
  Arms: Group 1; Group 3
Biological: Secretome — The topical secretome used is a hydrogel-based serum containing secretome components, including cytokines, growth factors, exosomes, microvesicles, and cell differentiation factors. The serum is formulated with a hydrogel base consisting of xanthan gum, sclerotium gum, 1% alginate, 2% glycerin, 1% caprylyl glycol, and 96% aqua. It is applied after cleansing the face with a facial cleanser, twice daily, in the morning and evening, for eight weeks
  Arms: Group 2; Group 3

SUMMARY:
Background: Acne vulgaris is a chronic inflammatory condition primarily caused by Cutibacterium acnes, which disrupts skin homeostasis, thereby triggering immune responses and sebum metabolism. Dysbiosis is an imbalances in the skin and gut microbiota identified as a significant factor contributing to acne progression. Standard therapy often rely on antibiotics, but the long-term use has increased antibiotic resistance, including in Indonesia. Consequently, alternative methods, such as probiotics and mesenchymal stromal cell (MSC) secretomes are gaining attention for immunomodulatory and regenerative properties. These novel therapies have shown promising results in modulating the skin and gut microbiota while reducing inflammation.

Study Design: A phase 2 double-blind randomized controlled trial was adopted using a parallel group design with four arms, namely: (1) standard therapy with oral probiotics and topical secretome (placebo), (2) standard therapy with oral probiotics (placebo) and topical secretome, (3) standard therapy with oral probiotics and topical secretome, and (4) standard therapy with oral probiotics (placebo) and topical secretome (placebo). Sixty-four mild to moderate acne vulgaris patients were randomly allocated to these groups. Interventions were administered over a period of 8 weeks, with outcomes measured at baseline and post-therapy. This study was conducted at Dermatology and Venereology Department of Bali Mandara General Hospital (RSBM). The primary outcome is the reduction of comedones and inflammatory lesions, assessed using the Yolov8 method. Secondary outcomes include gut and skin health parameters, such as tryptophan metabolites, collagen, pH, moisture, sebum levels, and IL-6, to explore the relationship between microbiome balance, skin condition, and inflammation in acne.

Discussion: In the context of increasing antibiotic resistance in Indonesia, where therapies often fail to produce sustainable clinical outcomes, this study showed the potential of combining probiotics and MSC secretomes as adjunctive therapies for acne vulgaris. Probiotics restored gut and skin microbiota balance, while MSC secretomes promoted immune modulation and tissue repair. The results of this study paved the way for innovative, non-antibiotic methods for acne management, addressing the need for sustainable and effective therapies amidst growing concerns over dysbiosis and antibiotic resistance.

DETAILED DESCRIPTION:
Acne cases have a very high number of visits to doctors, around 87%, especially in teenagers, which has implications for the psychological impact where long treatment with repeated inflammation for quite a long time can have the effect of reducing self-confidence and increasing stress. The therapy that is often given to Acne vulgaris is in the form of long-term topical antibiotics which can risk increasing the bacteria's resistance to antibiotics. Researchers are considering a new therapeutic approach in improving acne vulgaris by improving the balance of the microbiome through consuming oral probiotics so that it can reduce the development of C. acnes bacteria that cause acne and administering serum containing secretome to reduce inflammation/lesions in acne. As proof of the effect of the addition of this new therapy, research was carried out which required 64 research participants who met the criteria and consent from research participants was indicated by agreeing to take part in the research as outlined in the informed consent and research participants were asked to be involved until the research was completed. In research involving humans (participants) who experience mild to moderate acne as determined through examination by a dermatologist to determine the severity of the acne (seen from the total number of acne lesions or bumps), the patients included in the study had an age range of 13 - 45 years, and additional criteria such as: experiencing new acne lesions or bumps repeatedly in the last 6 months, willing to have flash facial images, and physically and mentally healthy. Research participants were given additional therapy from the therapy that should have been given by a doctor. The additional therapy was in the form of oral probiotics which had BPOM distribution permits and topical secretome in the form of facial serum. Participants will be divided into 4 groups randomly so that respondents are selected fairly and objectively. All drugs/test materials use natural ingredients which tend to be very safe with low side effects, oral probiotics have been reported in a few cases with diarrhea and secretome side effects with a very low possibility of skin redness, but to further increase safety, researchers will carry out a skin redness test first. first on the skin before being given the test material, and if changes occur such as loose stools and repeated bowel movements more than 3 times a day, the researchers have prepared medication as a preventive measure, and if it continues, it will be fully handled by the researchers. The development of new therapies, especially skin diseases, in this case Acne vulgaris, needs to be explored, one of which is through the microbiome approach and new regenerating medicine using stem cells (secretome). In this study, researchers want to prove that natural ingredient-based treatments, namely oral probiotics and topical secretome, can have the potential to improve acne vulgaris through measuring microbiome balance and severity, so in this study a clinical trial will be carried out to compare the effects of standard therapy (usual therapy) with additional oral probiotic therapy and topical secretome on its ability to increase clinical and microbiome improvement in moderate-severe Acne vulgaris patients through a double-blended open label Randomized Control Trial study.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 13 to 45 years
* diagnosed with acne vulgaris by a certified dermatologist, presenting with mild to moderate facial acne based on the lesion count criteria by Lehman et al. Mild acne is defined as having fewer than 20 comedones or fewer than 15 papular/pustular lesions, while moderate acne is characterized by 20-100 comedones and 20-50 papular/pustular lesions.
* must have experienced recurring new acne lesions in the past 6 months
* must be willing to comply with all protocol requirements
* must be willing to have standardized facial photograps taken using an imaging system
* must be able to follow study and adhere to a fixed schedule
* must have ability to provide inform concent for participation in the study
* must be generally healthy and in good mental condition.

Exclusion Criteria:

* pregnant patients
* subjects who have undergone hormonal acne treatment within six months prior to the study
* subjects who have taken oral isotretinoin within one month prior to the study.
* simultaneous participation in a different study conducted by an external research institution at the same testing site.
* inadequate language proficiency (both spoken and written)
* participation in the study under the influence of alcohol and/or drugs, as well as substance addiction
* severe diseases (cardiovascular, hepatic, renal, or pulmonary diseases, severe diabetes mellitus) or chronic infections (Hepatitis, HIV).
* immunodeficiency.
* current use of the following topical or systemic medications: corticosteroids, immunosuppressants, and antihistamines.
* skin conditions such as vitiligo, psoriasis, or atopic dermatitis.
* any other diseases or medications that may directly interfere with the study or pose a risk to the subject's health

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of comedones and inflammatory lesions | From enrollment to the end of treatment at 8 weeks
  The primary outcome measured in this study is the reduction in the number of comedones and/or inflammatory lesions (papules/pustules). This is assessed using the Yolov8 machine learning detection method, which enables accurate and objective quantification of comedones and lesions while also determining the severity of acne

SECONDARY OUTCOMES:
Tryptophan metabolites | From enrollment to the end of treatment at 8 weeks
  In the gut, tryptophan metabolites are measured using the ELISA method to assess the abundance of probiotic bacteria, specifically lactic acid bacteria such as Lactobacillus and Bifidobacterium
Inflammatory Response | From enrollment to the end of treatment at 8 weeks
  Inflammatory responses are assessed by measuring serum IL-6 levels, which serve as an indicator of systemic inflammation
Collagen Measurement | From enrollment to the end of treatment at 8 weeks
  collagen measurement use skin Elastometer
Moisture content | From enrollment to the end of treatment at 8 weeks
  Moisture content use skin hydrometer
Sebum levels | From enrollment to the end of treatment at 8 weeks
  Sebum levels use sebumeter
pH levels | From enrollment to the end of treatment at 8 weeks
  pH levels use pH meter to determine the balance of the skin microbiome

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Umum Daerah Bali Mandara, Denpasar, Bali, Indonesia